CLINICAL TRIAL: NCT04657523
Title: Pilot Study of On-Cart Liver Fat Quantification (LFQ) Feature to Assess Correlation With Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) Results
Brief Title: Ultrasound-Based Liver Fat Quantification (LFQ) Pilot Study
Acronym: LFQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: US-GIS-10481
Record Dates: First submitted 2020-11-20; First posted 2020-12-08 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2024-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis
Keywords: Liver Fat Quantification; Ultrasound; Liver Disease; Digestive System Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Digestive System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Investigational Ultrasound Imaging for Liver Fat Quantification (Experimental)
  Interventions: Device: Investigational Liver Fat Quantification Software

INTERVENTIONS:
Device: Investigational Liver Fat Quantification Software — All subjects enrolled in this study will undergo two abdominal ultrasound examinations using the investigational Liver Fat Quantification feature on the Philips EPIQ Ultrasound System. In addition, all subjects will also undergo one MRI-PDFF examination according to the clinical standard of care.

SUMMARY:
This clinical study will involve performing a series of medical imaging procedures of the abdomen using both ultrasound and MRI modalities in subjects at risk for or already diagnosed with Nonalcoholic Fatty Liver Disease (NAFLD). The primary objective of this clinical study is to evaluate the clinical feasibility of an investigational ultrasound technique for quantifying liver fat by comparing specific ultrasound-derived biomarkers with the liver fat percentage obtained from MRI Proton Density Fat Fraction (MRI-PDFF) measurements. All subjects enrolled in this study will undergo two investigational abdominal ultrasound examinations using the Philips EPIQ Ultrasound System and one MRI PDFF examination according to the clinical standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old and able to provide written informed consent
* Must attest to absent or minimal alcohol consumption (i.e. < 2 alcoholic beverages per day for women and < 3 alcoholic beverages per day for men, where an alcoholic beverage is defined as 12 oz. of regular beer, 5 oz. of wine, or 1.5 oz. of distilled spirits).
* Must be eligible for a standard abdominal ultrasound examination and standard non-contrast MRI examination.
* At least one of the following criteria must also be met: Overweight or obese (BMI ≥ 25); Diagnosed with Type 2 diabetes; Diagnosed with hypercholesterolemia; Diagnosed with or clinically suspected of having NAFLD/NASH

Exclusion Criteria:

* Evidence of moderate/heavy/binge alcohol consumption exceeding the thresholds above
* Evidence of hepatotoxicity
* History of chronic liver disease (e.g., viral, cholestatic, or autoimmune).
* Use of drugs associated with hepatic steatosis
* Subjects anticipated or planned to undergo any diagnostic or therapeutic intervention during enrollment period that, at discretion of the Investigator, may affect liver fat content
* Hepatic lesions that cannot be excluded from the imaging field during ultrasound LFQ data acquisition
* History of previous liver surgery or hepatic implants that, at the discretion of the Investigator, may adversely impact ultrasound or MRI image quality or the subject's eligibility to undergo ultrasound or MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony E. Samir, MD, Principal Investigator — Massachusetts General Hospital; Stephan Anderson, MD, Principal Investigator — Boston Medical Center; Richard G Barr, MD, PhD, Principal Investigator — Radiology Consultants, Inc
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Radiology Consultants, Inc, Boardman, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Started | 60 (60 participants)
Completed | 60 (60 participants)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 60 participants used for Baseline Characteristics
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 51
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Correlation of the Liver Fat Percentage Reported From MRI-PDFF With Measurements Hepatorenal Index (HRI) of Ultrasound Biomarkers for Liver Fat.
Description: For each biomarker per subject, multiple quantitative measurements were acquired on the same day by two different operators. The difference between the two operators was calculated at the subject level by averaging multiple measurements. To assess the correlation between measurements derived from the investigational LFQ feature and the 'clinical' MRI-PDFF fat fraction obtained from the subject's medical record. A higher HRI value indicates greater liver fat accumulation, which reflects a worse outcome, while a lower HRI suggests less hepatic fat and a better outcome.
Time Frame: Intra-procedural (1 day)
Population: Each enrolled subject underwent up to two ultrasound scans conducted by two different operators, resulting in a total of 119 non missing scans reviewed for this study. The primary outcome measure, the Hepatorenal Index, was calculated based on these scans. The hepatorenal index measurement from each ultrasound scan was reviewed.
Measure: Mean (Standard Deviation); unit: Hepatorenal Index
Units Other Than Participants: ultrasounds scans
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Number analyzed (ultrasounds scans) | 119
Hepatorenal Index | 1.6 (0.7)
Statistical Analysis 1: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the correlation between quantitative ultrasound biomarker "Hepatorenal Index (HRI)" derived from the investigational LFQ feature and the clinical MRI-PDFF fat fraction obtained from the subject's medical record. A higher HRI value indicates greater liver fat accumulation, which reflects a worse outcome, while a lower HRI suggests less hepatic fat and a better outcome; Test type: Other — Pearson correlation coefficient was calculated based on all measurements assuming independency; Pearson correlation coefficient = 0.5749
Statistical Analysis 2: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 1, analysis 1]; Test type: Other — Pearson correlation coefficient was calculated based on the subject level averages of multiple measurements; Pearson correlation coefficient = 0.6143
Statistical Analysis 3: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 1, analysis 1]; Test type: Other — To account for within subject variance in repeated measures by two different operators, a method with MIXED model for repeated measurements was used to estimate the correlation between two techniques with repeated measures. An unstructured covariance matrix was used; Mixed Model = 0.5944

2. Primary Outcome: Correlation of the Liver Fat Percentage Reported From MRI-PDFF With Measurements of Acoustic Attenuation (dB/cm/MHZ) Ultrasound Biomarker for Liver Fat.
Description: For each biomarker per subject, multiple quantitative measurements were acquired on the same day by two different operators. To assess the correlation between subject averaged measurements derived from the investigational LFQ feature and the 'clinical' MRI-PDFF fat fraction obtained from the subject's medical record.
  Correlation of each ultrasound biomarker with the liver fat percentage reported from MRI-PDFF is assessed independently to evaluate individual biomarker performance. A higher attenuation value indicates worse liver condition, while a lower attenuation value suggests better liver status.
Time Frame: Intra-procedural (1 day)
Population: Each enrolled subject underwent up to two ultrasound scans conducted by two different operators, resulting in a total of 120 scans reviewed for this study. The primary outcome measure, the Acoustic Attenuation (dB/cm/MHZ), was evaluated based on these scans.
Measure: Mean (Standard Deviation); unit: dB/cm/MHZ
Units Other Than Participants: Ultrasound scans
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Number analyzed (Ultrasound scans) | 120
dB/cm/MHZ | 1.0 (0.7)
Statistical Analysis 1: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the correlation between quantitative ultrasound biomarker "Acoustic attenuation " derived from the investigational LFQ feature and the clinical MRI-PDFF fat fraction obtained from the subject's medical record; Test type: Other — Pearson correlation coefficient was calculated based on all measurements assuming independency; Pearson correlation coefficient = 0.6824
Statistical Analysis 2: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 2, analysis 1]; Test type: Other — Pearson correlation coefficient was calculated based on the subject averages of multiple measurements; Pearson correlation coefficient = 0.7331
Statistical Analysis 3: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 3]; Correlation estimated from a mixed model = 0.7066

3. Primary Outcome: Correlation of the Liver Fat Percentage Reported From MRI-PDFF With Measurements of Tissue Stiffness (kPa) Ultrasound Biomarker for Liver Fat.
Description: For each biomarker per subject, multiple quantitative measurements were acquired on the same day by two different operators. To assess the correlation between subject averaged measurements derived from the investigational LFQ feature and the 'clinical' MRI-PDFF fat fraction obtained from the subject's medical record. This measured the MRI PDFF fat fraction used as the standard to evaluate the Tissue stiffness (kPa) measurements.
  Correlation of each ultrasound biomarker with the liver fat percentage reported from MRI-PDFF is assessed independently to evaluate individual biomarker performance.
Time Frame: Intra-procedural (1 day)
Population: Each enrolled subject underwent up to two ultrasound scans conducted by two different operators, resulting in a total of 120 scans reviewed for this study. The primary outcome measure, the Tissue Stiffness, was evaluated based on these scans.
Measure: Mean (Standard Deviation); unit: kPa
Units Other Than Participants: Ultrasound scans
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Number analyzed (Ultrasound scans) | 120
kPa | 5.9 (1.8)
Statistical Analysis 1: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the correlation between quantitative ultrasound biomarker "Tissue stiffness" derived from the investigational LFQ feature and the clinical MRI-PDFF fat fraction obtained from the subject's medical record; Test type: Other — Pearson correlation coefficient was calculated based on all observations assuming independency; Pearson correlation coefficient = -0.0539
Statistical Analysis 2: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 3, analysis 1]; Test type: Other — Pearson correlation coefficient was calculated based on the subject averages of multiple measurements; Pearson correlation coefficient = -0.0622
Statistical Analysis 3: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 3]; Correlation estimated from a mixed model = -0.0574

4. Secondary Outcome: To Evaluate the Same-day Inter-operator Variability for Investigating Biomarker "Hepatorenal Index (HRI)"
Description: To assess the difference in quantitative ultrasound biomarker measurements which acquired from the same subject on the same day by two different operators who have undergone standardized training for LFQ data acquisition. The difference between the two operators was calculated at the subject level by averaging multiple measurements. A higher HRI value indicates greater liver fat accumulation, which reflects a worse outcome, while a lower HRI suggests less hepatic fat and a better outcome.
Time Frame: Intra-procedural (1 day)
Population: The analysis included 119 ultrasound scans, performed by two different operators, from 60 enrolled participants. One participant scan was excluded due to missing Hepatorenal Index (HRI) data. The hepatorenal index measurement was calculated from each ultrasound scan and the difference between the two operators was reviewed.
Measure: Mean (Standard Deviation); unit: Hepatorenal Index
Units Other Than Participants: ultrasound scans
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Number analyzed (ultrasound scans) | 119
Hepatorenal Index | -0.1 (0.4)
Statistical Analysis 1: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the difference in quantitative ultrasound biomarker measurements which acquired from the same subject on the same day by two different operators who have undergone standardized training for LFQ data acquisition; Test type: Other — The Intra-class Correlation Coefficient (ICC) was calculated to test the same day inter-operator reliability. The estimated inter-operator correlation coefficient and the corresponding 95% confidence interval were reported; Intra-class Correlation Coefficient = 0.77, 95% CI 2-sided [0.64 to 0.86]

5. Secondary Outcome: To Evaluate the LFQ Data Acquisition Failure Rate for Investigating Biomarker "Hepatorenal Index (HRI)"
Description: To evaluate the LFQ data acquisition failure rate, the proportion of subjects who have at least one unacceptable image quality due to inadequate acoustic scanning windows, motion artifacts, or other technical limitations
Time Frame: Intra-procedural (1 day)
Population: To quantify the number of overall subjects with at least one unacceptable image quality
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Participants | 1
Statistical Analysis 1: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; To evaluate the LFQ data acquisition failure rate for the biomarker "Hepatorenal Index (HRI)"; Test type: Other — The proportion of subjects who have at least one unacceptable image quality due to inadequate acoustic scanning windows, motion artifacts, or other technical limitations and the associated 2-sided 95% binomial confidence intervals were calculated and summarized by each operator and overall; Proportion = 1.7, 95% CI 2-sided [0 to 4.9]

6. Secondary Outcome: To Evaluate the LFQ Data Acquisition Failure Rate for Investigating Biomarker Acoustic Attenuation (dB/cm/MHZ)
Description: as for outcome 5
Time Frame: Intra-procedural (1 day)
Population: 60 participants enrolled were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Participants | 0
Statistical Analysis 1: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; To evaluate the LFQ data acquisition failure rate for the biomarker "Acoustic attenuation (dB/cm/MHZ)"; Test type: Other — [test comment as in outcome 5, analysis 1]; Proportion = 0, 95% CI 2-sided [0 to 0]

7. Secondary Outcome: To Evaluate the LFQ Data Acquisition Failure Rate for Investigating Biomarker Tissue Stiffness (kPa)
Description: as for outcome 5
Time Frame: Intra-procedural (1 day)
Population: 60 participants enrolled were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Participants | 1
Statistical Analysis 1: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; To evaluate the LFQ data acquisition failure rate for the biomarker "Tissue stiffness (kPa)"; Test type: Other — [test comment as in outcome 5, analysis 1]; Proportion = 1.7, 95% CI 2-sided [0.0 to 4.9]

8. Secondary Outcome: To Evaluate the Same-day Inter-operator Variability for Investigating Biomarker Acoustic Attenuation (dB/cm/MHZ)
Description: To assess the difference in quantitative ultrasound biomarker measurements which acquired from the same subject on the same day by two different operators who have undergone standardized training for LFQ data acquisition.
  The difference between the two operators was calculated at the subject level by averaging multiple measurements.
Time Frame: Intra-procedural (1 day)
Population: The analysis included 120 ultrasound scans, performed by two different operators, from 60 enrolled participants. The Acoustic attenuation (dB/cm/MHZ) calculated from each ultrasound scan and the difference between the two operators was reviewed.
Measure: Mean (Standard Deviation); unit: dB/cm/MHZ
Units Other Than Participants: ultrasound scans
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Number analyzed (ultrasound scans) | 120
dB/cm/MHZ | 0.0 (0.1)
Statistical Analysis 1: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; To assess the difference in quantitative ultrasound biomarker Acoustic attenuation measurements which acquired from the same subject on the same day by two different operators who have undergone standardized training for LFQ data acquisition; Test type: Other — The Intra-class Correlation Coefficient (ICC) was calculated to assess the same day inter-operator reliability. The estimated inter-operator correlation coefficient and the corresponding 95% confidence interval were reported; Intra-class Correlation Coefficient = 0.74, 95% CI 2-sided [0.60 to 0.84]

9. Secondary Outcome: To Evaluate the Same-day Inter-operator Variability for Investigating Biomarker Tissue Stiffness (kPa)
Description: as for outcome 8
Time Frame: Intra-procedural (1 day)
Population: The analysis included 120 ultrasound scans, performed by two different operators, from 60 enrolled participants. The Tissue stiffness (kPa) was calculated from each ultrasound scan and the difference between the two operators was reviewed.
Measure: Mean (Standard Deviation); unit: Tissue stiffness (kPa)
Units Other Than Participants: ultrasound scans
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
Number analyzed (Participants) | 60
Number analyzed (ultrasound scans) | 120
Tissue stiffness (kPa) | 0.1 (1.9)
Statistical Analysis 1: Comparison: Investigational Ultrasound Imaging for Liver Fat Quantification; [analysis description as in outcome 4, analysis 1]; Test type: Other — The Intra-class Correlation Coefficient (ICC) was calculated to test the inter-operator reliability. The estimated inter-operator correlation coefficient and the corresponding 95% confidence interval were reported; Intra-class Correlation Coefficient = 0.51, 95% CI 2-sided [0.30 to 0.67]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: There are no significant Anticipated Adverse Events and Anticipated Adverse Device Effects associated with this clinical study because the investigational procedure is limited to noninvasive diagnostic ultrasound imaging of the abdomen using the investigational LFQ software.
Arm/Group | Investigational Ultrasound Imaging for Liver Fat Quantification
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT04657523/Prot_SAP_001.pdf